CLINICAL TRIAL: NCT05810246
Title: 68Ga-NY104 PET/CT and Conventional Imaging in Patients With Von Hippel-Lindau Disease: a Prospective, Single-center, Single-arm, Comparative Imaging Study
Brief Title: 68Ga-NY104 PET/CT in Von Hippel-Lindau Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYCOV
Record Dates: First submitted 2023-03-09; First posted 2023-04-12 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Von Hippel-Lindau Disease
MeSH Terms: conditions — von Hippel-Lindau Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic imaging arm (Experimental): 68Ga-NY104 PET/CT Contrast-enhanced MRI of the brain and contrast-enhanced CT of abdomen and pelvis 68Ga-NODAGA-LM3 PET/CT (exploratory)
  Interventions: Diagnostic Test: 68Ga-NY104 PET/CT Contrast-enhanced MRI of the brain and contrast-enhanced CT of abdomen and pelvis) 68Ga-NODAGA-LM3 PET/CT (exploratory)

INTERVENTIONS:
Diagnostic Test: 68Ga-NY104 PET/CT Contrast-enhanced MRI of the brain and contrast-enhanced CT of abdomen and pelvis) 68Ga-NODAGA-LM3 PET/CT (exploratory) — 68Ga-NY104 PET/CT is expected to be completed within 21 days following screening. Participants will be administered a single, intravenous bolus of 68Ga-NY104 (1.8-2.2 MBq per kilogram bodyweight). PET/CT scanning will occur at 45 -75 minutes following injection of 68Ga-NY104.
  Conventional imaging should be performed within one month from 68Ga-NY104 PET/CT. It includes contrast-enhanced MRI of brain and contrast-enhanced CT of abdomen and pelvis.
  68Ga-NODAGA-LM3 PET/CT is optional in patients with evidence of or in suspicion of pheochromocytoma, paraganglioma, or pancreatic neuroendocrine tumor. They are encouraged to undergo exploratory 68Ga-NODAGA-LM3 PET/CT for better evaluation of neuroendocrine tumors. The decision, however, is up to the participants. 68Ga-NODAGA-LM3 PET/CT should be performed within one month after 68Ga-NY104 PET/CT. The details of 68Ga-NODAGA-LM3 PET/CT are similar to 68Ga-NY104 PET/CT.

SUMMARY:
This is a prospective, single-center, single-arm, diagnostic phase 2 study in patients with von Hippel-Lindau disease. VHL disease is a rare syndrome characterized by VHL gene mutation and HIF activation. Although genetic testing is available, the manifestations of the syndrome are protean; therefore, imaging plays a crucial role in the identification of abnormalities and subsequent follow-up of lesions. For now, conventional imaging serves as the main radiologic modality in the characterization of VHL disease. In this study, we aim to evaluate the sensitivity of 68Ga-NY104 PET/CT in patients with VHL disease. 68Ga-NY104 is a novel small molecule PET tracer targeting carbonic anhydrase IX, which is a down-streaming target of HIF and overexpressed in HIF activation. 68Ga-NY104 PET/CT is likely to function as a sensitive imaging tool to identify VHL-related tumors and to impact patient management if additional lesions are identified.

The hypotheses of this study are that

* 68Ga-NY104 PET/CT can be used as an effective imaging modality in VHL syndrome with high sensitivity
* 68Ga-NY104 PET/CT may detect lesions that are missed on conventional imaging and can result in management impact.

A total of 19 patients will be recruited at Peking Union Medical College Hospital. As an exploratory end-point, a 68Ga-NODAGA-LM3 PET/CT sub-study will be performed in patients with evidence of neuroendocrine tumors.

DETAILED DESCRIPTION:
Hypothesis

The hypotheses of this study are that

* 68Ga-NY104 PET/CT can be used as an effective imaging modality in VHL syndrome with high sensitivity
* 68Ga-NY104 PET/CT may detect lesions that are missed on conventional imaging and can result in management impact.

Objectives

Primary objective 1. To determine the sensitivity of 68Ga-NY104 PET/CT using conventional imaging as reference.

Secondary objectives

1. To determine the incremental management impact of 68Ga-NY104 PET/CT
2. To assess the interobserver agreement of 68Ga-NY104 PET/CT by comparing the two blinded independent readings

Exploratory objective

1. To compare the per-patient, per-region, and per-lesion sensitivity of 68Ga-NY104 PET/CT to 68Ga-NODAGA-LM3 PET/CT in an exploratory endpoint

Endpoints

Primary endpoint 1. Per-patient, per-region, and per-lesion positive rate of 68Ga-NY104 using conventional imaging as ground truth.

Secondary endpoints

1. Incremental impact of 68Ga-NY104 PET/CT on choice of management, defined as a decision to alter the original plan of treatment (based on conventional imaging) after considering the result of 68Ga-NY104 PET/CT (Impact is categorized as high, medium, low or no incremental impact.)
2. Observer agreement in interpretation of 68Ga-NY104 PET/CT between the two independent nuclear medicine readers.

Exploratory endpoints

1. Per-patient, per-region, and per-lesion positive rate of 68Ga-NODAGA-LM3 using conventional imaging as ground truth.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of VHL disease, according to 2022 CSCO guideline, if any one of the following criteria is met: germline VHL alteration, family history of VHL syndrome as well as presence of at least one VHL related tumor (including hemangioblastoma, clear cell renal cell tumor, pheochromocytoma, paraganglioma, pancreatic neuroendocrine tumor, etc.), two or more hemangioblastoma, hemangioblastoma and pheochromocytoma, hemangioblastoma and clear cell renal cell tumor.
2. Age ≥ 18 y
3. Written informed consent provided for participation in the trial
4. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. Patients on VEGF TKI treatment < 1 week before 68Ga-NY104 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC and is expected to have the same effect on 68Ga-NY104. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NY104 PET/CT is required.
2. Patients on HIF antagonist treatment < 3 months before 68Ga-NY104 PET/CT. CA9, which encodes carbonic anhydrase IX (CAIX), is one of the genes most strongly upregulated by HIF-1. HIF antagonist, such as Belzutifan, might affect the expression of CAIX and thus the binding of 68Ga-NY104 to tumor. Withdraw of at least 3 months is required for HIF antagonist.
3. Patients with known allergic reaction to CT or MR contrast medium.
4. Patients with renal dysfunction
5. Pregnancy or breastfeeding.
6. Severe claustrophobia.
7. If the patient will undergo an exploratory 68Ga-NODGA-LM3 PET/CT and is on cold somatostatin analogue (such as Octreotide and Lanreotide), the 68Ga-NODGA-LM3 should be injected at least 24 hours after cold somatostatin analogue injection. Patients violating this criteria will not be able to attend the exploratory 68Ga-NODGA-LM3 PET/CT study but will still be considered eligible for the main study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Binary reading of lesions identified on 68Ga-NY104 PET/CT | From study completion to 1 month after completion
  Define lesion as PET positive or PET negative lsion
The number of (68Ga-NY104) PET positive lesions | From study completion to 1 month after completion
  Count the number of lesions (if more than 10, record it as >10)
The number of (68Ga-NY104) PET positive regions | From study completion to 1 month after completion
  Any region with at least one (68Ga-NY104) PET positive lesion is considered (68Ga-NY104) PET positive VHL-related region
The number of (68Ga-NY104) PET positive patients | From study completion to 1 month after completion
  Any patient with at least one (68Ga-NY104) PET positive lesion is considered (68Ga-NY104) PET positive VHL-related patient
Scoring of lesions identified on conventional imaging as very unlikely / unlikely / indeterminate / likely / very likely (score 1-5) | From study completion to 1 month after completion
  The likelihood of VHL-related neoplasm will be rated combining all imaging features available, including enhancement pattern, typical location, and solitary or multicentric or bilateral distribution.
The number of conventional imaging positive lesions | From study completion to 1 month after completion
  Count the number of lesions (if more than 10, record it as >10)
The number of conventional imaging positive regions | From study completion to 1 month after completion
  Any region with at least one conventional-imaging positive VHL-related lesion is considered conventional-imaging positive VHL-related region
The number of conventional imaging positive patients | From study completion to 1 month after completion
  Any patient with at least one conventional-imaging positive VHL-related lesion is considered conventional-imaging positive VHL-related patient

SECONDARY OUTCOMES:
The intent of initial management plan (Plan 1) based on conventional imaging | From study completion to 1 month after completion
  Management plan intent (curative, palliative or surveillance): it should be noted that the curative intent in the present study could be organ specific. For example, if the patient has non-symptomatic CNS hemangioblastomas and a solitary renal cell carcinoma, the intent to resect the renal cell carcinoma should be defined as "curative" even if the CNS hemangioblastomas are left undealt with.
The intent of post-PET management plan (Plan 2) based on all information available, including the results of conventional imaging, 68Ga-NY104 PET/CT, and additional confirmatory studies. | From study completion to 1 month after completion
  Management plan intent (curative, palliative or surveillance): it should be noted that the curative intent in the present study could be organ specific. For example, if the patient has non-symptomatic CNS hemangioblastomas and a solitary renal cell carcinoma, the intent to resect the renal cell carcinoma should be defined as "curative" even if the CNS hemangioblastomas are left undealt with.
The specified management plan of initial management plan (Plan 1) based on conventional imaging | From study completion to 1 month after completion
  Specified management plan for each patient including details of surgery or medical treatment or active surveillance. For surgery, this will include type of surgery (e.g., partial nephrectomy or radical nephrectomy, with / without lymph node dissection). For medical treatment, this will include the regimen, dose, and frequency of the treatment plan. For active surveillance, this will include the type and frequency of modality.
The specified management plan of post-PET management plan (Plan 2) based on all information available, including the results of conventional imaging, 68Ga-NY104 PET/CT, and additional confirmatory studies. | From study completion to 1 month after completion
  Specified management plan for each patient including details of surgery or medical treatment or active surveillance. For surgery, this will include type of surgery (e.g., partial nephrectomy or radical nephrectomy, with / without lymph node dissection). For medical treatment, this will include the regimen, dose, and frequency of the treatment plan. For active surveillance, this will include the type and frequency of modality.

OTHER OUTCOMES:
Binary reading of lesions identified on 68Ga-NODAGA-LM3 PET/CT as PET positive lesions or PET negative lesions | From study completion to 1 month after completion
  Define lesion as PET positive or PET negative lsion
The number of (68Ga-NODAGA-LM3) PET positive lesions | From study completion to 1 month after completion
  Count the number of lesions (if more than 10, record it as >10)
The number of (68Ga-NODAGA-LM3) PET positive regions | From study completion to 1 month after completion
  Any region with at least one (68Ga-NODAGA-LM3) PET positive lesion is considered (68Ga-NODAGA-LM3) PET positive VHL-related region
The number of (68Ga-NODAGA-LM3) PET positive patients | From study completion to 1 month after completion
  Any patient with at least one (68Ga-NODAGA-LM3) PET positive lesion is considered (68Ga-NODAGA-LM3) PET positive VHL-related patient

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 2 years after the publication of the main results
Access Criteria: No limit.